CLINICAL TRIAL: NCT04363814
Title: A Prospective, Open-label, Randomized Pilot Study (Including a Control Group) of BACTEK-R (MV130), Administered Sublingually to Assess the Clinical Impact in Subjects With Mild Pneumonia Due to COVID-19
Brief Title: Clinical Impact of BACTEK-R in Subject With Mild Pneumonia Due to COVID-19 Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Inmunotek S.L. (Industry)
Collaborators: BioClever 2005 S.L. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MV130-SLG-35
Record Dates: First submitted 2020-04-19; First posted 2020-04-27 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bactek-R (Experimental): Subject included in the experimental group will receive Bactek- R.The dose consists on 3 spray puff every 6 hours for 2 weeks.
  Interventions: Biological: Bactek-R
- Control (No Intervention): Subject included in the control group will receive standard therapy for COVID-19.

INTERVENTIONS:
Biological: Bactek-R — BACTEK-R is a bacterial preparation that contains a mixture of Gram + and Gram - inactivated bacteria at the concentration of 300 FTU / mL (approx. 10^9 bacteria / mL)
  Arms: Bactek-R

SUMMARY:
The purpose of the study is to confirm if BACTEK-R (MV130) provides clinical benefit in subject with mild pneumonia (CURB-65≤2) by COVID-19 admitted to the Hospital.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized pilot study to evaluate the efficacy and safety of BACTEK-R (MV130) in subject with mild pneumonia due to COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. - Subjects who voluntarily sign informed consent forms
2. - Both genders.
3. - Subjects aged between 18 and 70 years.
4. -Subjects capable of complying with the treatment
5. - Subjects admitted to hospital with non-severe pneumonia (CURB-65≤2) by COVID-19
6. - Confirmatory test for COVID-19 infection

Exclusion Criteria:

1. - Subjects who has not signed informed consent forms
2. - Subjects included in another clinical trial.
3. - Subjects under treatment with immunosuppressants.
4. - Subjects in treatment with another type of immunotherapy.
5. - Subjects who are or have been undergoing treatment with metformin.
6. - Subjects who are or have been treated with statins.
7. - Subjects who are or have been under treatment with sertraline.
8. - Pregnant women.
9. - Subjects who cannot offer cooperation and / or have serious psychiatric disorders.
10. -Subjects who are allergic to any of the components of BACTEK-R (MV130).
11. - Subjects with pathologies described in the Charlson index

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical recovery | 2 weeks
  Number of subjects presenting a improvement in their clinical condition from day 1 to 14 that lead their hospital discharged. Based on the measure of the secondary outcomes.
Clinical worsening | 2 weeks
  Number of subjects presenting a worsening in their clinical condition from day 1 to 14 that leads to their admission to the intensive care unit or their death. Based on the measure of the secondary outcomes.

SECONDARY OUTCOMES:
Clinical severity | 2 weeks
  Symptom (fever, cough, dyspnea, myalgia, diarrhea and so on) will be daily record and classified as mild, moderate, severe.
Time to symptoms remission | 2 weeks
  Time of reduction or disappearance of the symptoms
Medication Use | 2 weeks
  Record of all the medication administered to the subject
Hospitalization time | 2 weeks
  Time from the subject's admission to the coronavirus unit until discharge
Blood routine test | Days 1 and 7
  Blood routine test will be carried out days 1 and 7
Heart rate | 2 weeks
  Heart rate will be followed everyday during time frame
Blood pressure | 2 weeks
  Blood pressure will be followed everyday during time frame
Cardiac auscultation | 2 weeks
  Cardiac auscultation will be recorded everyday during time frame
Oxygen saturation | 2 weeks
  Blood oxygen saturation will be followed everyday during time frame
Adverse events | 2 weeks
  Adverse events during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Martín Medrano, MD, Principal Investigator; Nicolas Batlle, MD, Principal Investigator; Raymundo Hernández, Principal Investigator; Natalia García, Principal Investigator; M. Polanco, Principal Investigator; Guillermo Ángeles, Study Director
Locations (1):
- Hospital Metropolitano Santiago, Santiago de los Caballeros, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cirauqui C, Benito-Villalvilla C, Sanchez-Ramon S, Sirvent S, Diez-Rivero CM, Conejero L, Brandi P, Hernandez-Cillero L, Ochoa JL, Perez-Villamil B, Sancho D, Subiza JL, Palomares O. Human dendritic cells activated with MV130 induce Th1, Th17 and IL-10 responses via RIPK2 and MyD88 signalling pathways. Eur J Immunol. 2018 Jan;48(1):180-193. doi: 10.1002/eji.201747024. Epub 2017 Sep 14. PMID 28799230
- [Background] Esposito S, Soto-Martinez ME, Feleszko W, Jones MH, Shen KL, Schaad UB. Nonspecific immunomodulators for recurrent respiratory tract infections, wheezing and asthma in children: a systematic review of mechanistic and clinical evidence. Curr Opin Allergy Clin Immunol. 2018 Jun;18(3):198-209. doi: 10.1097/ACI.0000000000000433. PMID 29561355
- [Background] Sanchez-Ramon S, Perez de Diego R, Dieli-Crimi R, Subiza JL. Extending the clinical horizons of mucosal bacterial vaccines: current evidence and future prospects. Curr Drug Targets. 2014;15(12):1132-43. doi: 10.2174/1389450115666141020160705. PMID 25330031
- [Background] Tejera-Alhambra M, Palomares O, Perez de Diego R, Diaz-Lezcano I, Sanchez-Ramon S. New Biological Insights in the Immunomodulatory Effects of Mucosal Polybacterial Vaccines in Clinical Practice. Curr Pharm Des. 2016;22(41):6283-6293. doi: 10.2174/1381612822666160829143129. PMID 27573928
- [Background] Alecsandru D, Valor L, Sanchez-Ramon S, Gil J, Carbone J, Navarro J, Rodriguez J, Rodriguez-Sainz C, Fernandez-Cruz E. Sublingual therapeutic immunization with a polyvalent bacterial preparation in patients with recurrent respiratory infections: immunomodulatory effect on antigen-specific memory CD4+ T cells and impact on clinical outcome. Clin Exp Immunol. 2011 Apr;164(1):100-7. doi: 10.1111/j.1365-2249.2011.04320.x. PMID 21391984
- [Background] Sanchez Ramon S, Manzanares M, Candelas G. MUCOSAL anti-infections vaccines: Beyond conventional vaccines. Reumatol Clin (Engl Ed). 2020 Jan-Feb;16(1):49-55. doi: 10.1016/j.reuma.2018.10.012. Epub 2018 Dec 7. English, Spanish. PMID 30527360
- [Background] Sanchez-Ramon S, Conejero L, Netea MG, Sancho D, Palomares O, Subiza JL. Trained Immunity-Based Vaccines: A New Paradigm for the Development of Broad-Spectrum Anti-infectious Formulations. Front Immunol. 2018 Dec 17;9:2936. doi: 10.3389/fimmu.2018.02936. eCollection 2018. PMID 30619296
- [Background] Del-Rio-Navarro BE, Espinosa Rosales F, Flenady V, Sienra-Monge JJ. Immunostimulants for preventing respiratory tract infection in children. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD004974. doi: 10.1002/14651858.CD004974.pub2. PMID 17054227
- [Background] Lusuardi M. Challenging mucosal immunity with bacterial extracts to prevent respiratory infections: an old therapy revisited. Monaldi Arch Chest Dis. 2004 Jan-Mar;61(1):4-5. No abstract available. PMID 15366329
- [Background] Garcia Gonzalez LA, Arrutia Diez F. Mucosal bacterial immunotherapy with MV130 highly reduces the need of tonsillectomy in adults with recurrent tonsillitis. Hum Vaccin Immunother. 2019;15(9):2150-2153. doi: 10.1080/21645515.2019.1581537. Epub 2019 Apr 17. PMID 30779677
- [Background] Molero-Abraham M, Sanchez-Trincado JL, Gomez-Perosanz M, Torres-Gomez A, Subiza JL, Lafuente EM, Reche PA. Human Oral Epithelial Cells Impair Bacteria-Mediated Maturation of Dendritic Cells and Render T Cells Unresponsive to Stimulation. Front Immunol. 2019 Jun 28;10:1434. doi: 10.3389/fimmu.2019.01434. eCollection 2019. PMID 31316504
- [Background] Randomised double-blind placebo-controlled, parallel, multi-centre clinical trial of sublingual bacterial vaccine in children with recurrent bronchospasm (wheezing attacks) for the evaluation of efficacy, security and clinical impact.